CLINICAL TRIAL: NCT00437151
Title: An Analysis of Adherence and Associated Factors in Subjects Undergoing Differin® Gel, 0.1% Treatment of Moderate to Severe Acne Vulgaris.
Brief Title: Analysis of Adherence & Associated Factors in Teenagers Undergoing Treatment of Acne Vulgaris With Differin® Gel 0.1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10022
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Voice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): More frequent than normal office visits
  Interventions: Other: More frequent than normal office visits
- 2 (Active Comparator): Electronic reminders (voice, e-mail, text messages)
  Interventions: Other: Electronic reminders (voice, e-mail, text messages)
- 3 (Active Comparator): Parental involvement / intervention reminders
  Interventions: Other: Parenteral involvement / intervention reminders
- 4 (Active Comparator): No intervention or reminders
  Interventions: Other: No intervention or reminders

INTERVENTIONS:
Other: More frequent than normal office visits — Mode of patient reminder
  Arms: 1
Other: Electronic reminders (voice, e-mail, text messages) — Mode of patient reminder
  Arms: 2
Other: Parenteral involvement / intervention reminders — Mode of patient reminder
  Arms: 3
Other: No intervention or reminders — Mode of patient reminder
  Arms: 4

SUMMARY:
The primary objective of this study is to investigate potential differences in treatment adherence by teenagers among four interventions during treatment for acne.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent subjects with a diagnosis of moderate to severe Acne vulgaris

Exclusion Criteria:

* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or severe acne requiring more than topical treatment (e.g. oral isotretinoin)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy - Percent adherence calculated from MEMS Caps readings | 12 weeks

SECONDARY OUTCOMES:
Efficacy - lesion counts; percent adherence as calculated by product weights and by Subject's Diary; Global Severity Assessment; Global Assessment of Improvement; Subject questionnaire | 12 weeks
Safety - tolerability and adverse event reporting | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma Laboratories, LP
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States